CLINICAL TRIAL: NCT06124365
Title: Effect of Adding Shock Wave Therapy to Core Stability Exercises in Treatment of Postpartum Sacroiliac Joint Pain: A Single-blinded, Randomized Controlled Trial.
Brief Title: Shock Wave and Core Exercises for Postpartum Sacroiliac Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Postpartum sacroiliac pain
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Postpartum Sacroiliac Joint Pain
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: Shock wave therapy and core stability exercises
- Control group (Active Comparator)
  Interventions: Other: core stability exercises only

INTERVENTIONS:
Other: Shock wave therapy and core stability exercises — 20 post-partum women with SIJP will be treated by ESWT once weekly combined with core stability exercises 3 times per week for 6 weeks.
  Arms: study group
Other: core stability exercises only — 20 post-partum women with SIJP will be treated by core stability exercises 3 times per week for 6 weeks.
  Arms: Control group

SUMMARY:
Despite the high popularity and novelty of shock wave therapy (SWT), it is surprising that just one study has examined the effect of SWT on patients with SIJD and their functional ability following treatment by using subjective assessment tools like numeric rating scale (NRS) and limited by its small sample size and lack of long-term follow-up. Therefore, the present study is expected to contribute to the body of knowledge by exploring the effect of adding SWT to core stability exercises in the management of postpartum sacroiliac joint pain.

ELIGIBILITY:
Inclusion Criteria:

* post-partum women diagnosed with SIJP with limitation of its movement referred from the orthopedist.
* Age is between 25-35 years old.
* Their body mass index will be ranged from 25-35 kg/m2.

Exclusion Criteria:

Patients who have one of the following criteria will be excluded from the study:

* Previous spinal surgery.
* Medical diagnosis other than SIJ dysfunction.
* Patients who had any other spine disorders.
* Patients who had leg length discrepancies.
* Patients with congenital postural deformities.
* Patients with spinal cord injury or acute or unstable neurological signs.
* Patients with cauda equina symptoms related to the spine including changes in bowel or bladder control and perineal sensation.
* Patients with lumber intervertebral disc, spondylosis, lumbar canal stenosis and spondylolysthesis.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Sacroiliac joint pain intensity | change from base line at 6 weeks.
  Sacroiliac joint pain intensity will be measured by visual analogue scale
pain pressure threshold | change from base line at 6 weeks.
  pain pressure threshold will be measured by pressure algometer
functional disability | change from base line at 6 weeks
  functional disability will be measured by Oswestry disability index

SECONDARY OUTCOMES:
quality of life | change from base line at 6 weeks.
  quality of life will be measured by the standard quality of life assessment tool which is known as the short-form SF 36 tool